CLINICAL TRIAL: NCT02916758
Title: Let's Go: Promoting Community Mobility for Wellness in Older Adults in Urban Environments
Brief Title: Promoting Community Mobility for Wellness in Older Adults in Urban Environments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kean University (Other)
Responsible Party: Principal Investigator, Claire M. Mulry, OTD, OTR, CAPS, Assistant Professor, Kean University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Kean-1001
Record Dates: First submitted 2016-09-22; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
Keywords: older adults; community mobility; wellness; isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Let's Go Community Mobility Program (Experimental): Participation in 4 week program
  Interventions: Other: Let's Go Community Mobility Program

INTERVENTIONS:
Other: Let's Go Community Mobility Program — Four week multi-modal education and experiential program to improve community mobilty

SUMMARY:
This study evaluates the program outcomes of the Let's Go program. The standardized community mobility program employs multi-modal group and individual sessions to facilitate wellness in older adults.

DETAILED DESCRIPTION:
This study examines the outcomes of Let's Go, a standardized community mobility program which employs group and individual sessions of education, peer interaction, engagement in meaningful occupations, and self-reflections to help individuals understand the importance of community participation and its relationship to well-being. Program outcomes explored include increased confidence in community mobility, increased autonomy outdoors, social life and relationships, frequency of community trips, and decreased social isolation.

ELIGIBILITY:
Inclusion Criteria:

1. Community dwelling individual
2. Report desire to learn about community mobility options
3. Able to participate in group education sessions (
4. Able to attend during a 45 minute session
5. Independent mobility in community with or without an assistive device.

Exclusion Criteria:

1. Individual lives in Long Term Care facility
2. Aphasia
3. Individual has impaired cognition demonstrated by MoCA exam score ≤ 17
4. Individual is unable to stay awake for entire group session
5. Individual acts out (yelling, monopolizes, motor restlessness or agitation) in group setting.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in Impact on Participation and Autonomy Questionnaire-Autonomy Outdoors Sub scale | Baseline, 4 weeks (program end), 6 month follow up
  The IPAQ measures an individual's perception of the impact of chronic disability on participation, has good responsiveness and its content, construct, and discriminant validity as well as internal consistency are deemed adequate and verified by Rasch analysis (Magasi & Post, 2010). The content validity of the autonomy outdoors subscale (α = .81) and social life and relationships scale (α = .86) are strong. Internal reliability of the IPAQ on all subscales is high (all Cronbach's alphas >0.8). The individual items on the AO subscale have a test-retest reliability ranging from .69 to .84 and those on the SL subscale ranged from Kw = .71 to .77 (Cardol et al., 1999, Sibley et al., 2006).
Change in Impact on Participation and Autonomy Questionnaire- Social Life and Relationships Sub scale | Baseline, 4 weeks (program end), 6 month follow up
  The IPAQ measures an individual's perception of the impact of chronic disability on participation, has good responsiveness and its content, construct, and discriminant validity as well as internal consistency are deemed adequate and verified by Rasch analysis (Magasi & Post, 2010). The content validity of the autonomy outdoors subscale (α = .81) and social life and relationships scale (α = .86) are strong. Internal reliability of the IPAQ on all subscales is high (all Cronbach's alphas >0.8). The individual items on the AO subscale have a test-retest reliability ranging from .69 to .84 and those on the SL subscale ranged from Kw = .71 to .77 (Cardol et al., 1999, Sibley et al., 2006).
Change in Frequency of community trips per month | Baseline, 4 weeks (program end), 6 month follow up
  A Participant Survey was developed by the Primary Investigator in which participants self reported the frequency of community trips in the past 30 days
Change in Confidence in community mobility | Baseline, 4 weeks (program end), 6 month follow up
  A Participant Survey was developed by the Primary Investigator in which participants self reported their confidence in community mobility on a Likert Scale
Change in Self report of feelings of isolation | Baseline, 4 weeks (program end), 6 month follow up
  A Participant Survey was developed by the Primary Investigator in which participants self reported their feeling of isolation on a Likert Scale

CONTACTS AND LOCATIONS:
Overall Officials: Claire M Mulry, Principal Investigator — Kean University
Locations (1):
- Kean University, Union, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Data files will be uploaded for review

REFERENCES:
- [Background] Mulry, C. M. & Piersol, C. V. (2014). The Let's Go program for community participation: A feasibility study. Physical & Occupational Therapy in Geriatrics, 32(3). doi:10.3109/02703181.2014.932316
- [Derived] Mulry CM, Papetti C, De Martinis J, Ravinsky M. Facilitating Wellness in Urban-Dwelling, Low-Income Older Adults Through Community Mobility: A Mixed-Methods Study. Am J Occup Ther. 2017 Jul/Aug;71(4):7104190030p1-7104190030p7. doi: 10.5014/ajot.2017.025494. PMID 28661382
- Available data/document: Individual Participant Data Set — http://grad.kean.edu/ot/faculty — Please contact cmulry@kean.edu to request the data set